CLINICAL TRIAL: NCT04787341
Title: Randomized Phase II Study of Panitumumab Rechallenge Followed by Regorafenib Versus the Reverse Sequence in RAS and BRAF Wild-type Chemorefractory Mestastatic Colorectal Cancer Patients
Brief Title: PAnitumumab REchallenge Followed by REgorafenib Versus the Reverse Sequence
Acronym: PARERE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Collaborators: Bayer (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUDRACT 2019-002834-35
Record Dates: First submitted 2021-02-24; First posted 2021-03-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib; Panitumumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Panitumumab followed by Regorafenib (Active Comparator)
  Interventions: Drug: Panitumumab
- Regorafenib followed by Panitumumab (Experimental)
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — regorafenib administered until progression, unacceptable toxicity or patient's refusal followed after progression by panitumumab until further progression, unacceptable toxicity or patient's refusal in RAS and BRAF wt mCRC patients with the following characteristics:
  1. previous treatment with, or not considered candidates for, fluoropyrimidine, oxaliplatin, irinotecan and anti-angiogenic agent (bevacizumab or aflibercept);
  2. RECIST response or stable disease lasting at least 6 months to a previous first-line anti-EGFR-based treatment;
  3. RAS and BRAF wt ct-DNA at the time of screening.
  Other Names: panitumumab
  Arms: Regorafenib followed by Panitumumab
Drug: Panitumumab — panitumumab administered until progression, unacceptable toxicity or patient's refusal followed after progression by regorafenib until further progression, unacceptable toxicity or patient's refusal in RAS and BRAF wt mCRC patients with the following characteristics:
  1. previous treatment with, or not considered candidates for, fluoropyrimidine, oxaliplatin, irinotecan and anti-angiogenic agent (bevacizumab or aflibercept);
  2. RECIST response or stable disease lasting at least 6 months to a previous first-line anti-EGFR-based treatment;
  3. RAS and BRAF wt ct-DNA at the time of screening.
  Other Names: regorafenib
  Arms: Panitumumab followed by Regorafenib

SUMMARY:
The association of doublet chemotherapy (FOLFOX and FOLFIRI) and anti-EGFR-moAbs (panitumumab or cetuximab) is a standard option for the first-line treatment of unresectable RAS and BRAF wt mCRC patients, especially with left-sided primary tumour.

In RAS wt mCRC patients refractory to chemotherapy and anti-EGFR naive, the standard treatment sequence is an anti-EGFR-based therapy (panitumumab or cetuximab +/- irinotecan) followed by regorafenib.

In a phase II randomized Japanese study named REVERCE, a higher OS was reported in favour of an experimental strategy of regorafenib followed at progression by cetuximab +/- irinotecan compared with the reverse standard sequence in chemorefractory and anti-EGFR-naïve, RAS wt mCRC patients.

However, the limitations of the REVERCE study (phase II trial with a premature conclusion for poor accrual) do not allow us to draw definitive conclusions. In addition, nowadays, patients candidates to an anti-EGFR-based treatment, receive anti-EGFRMoAbs in earlier lines of therapy thus affecting the translation of these results in the current clinical practice.

Retrospective analyses and a phase II single-arm trial showed promising activity of anti-EGFR rechallenge in patients who previously achieved benefit from a first-line anti- EGFR-based treatment and not bearing RAS mutation on ct-DNA at the rechallenge baseline.

Based on these considerations, the Investigators designed the present phase II randomized study of panitumumab followed at progression by regorafenib versus the reverse sequence in RAS and BRAF wt mCRC patients with the following characteristics:

1. previous treatment with, or not considered candidates for, fluoropyrimidine, oxaliplatin, irinotecan and an anti-angiogenic agent (bevacizumab or aflibercept);
2. RECIST response or stable disease lasting at least 6 months to a previous first-line anti-EGFR-based treatment;
3. RAS and BRAF wt ct-DNA at the time of screening. The aim of this study is to compare the two sequences in a Caucasian population of patients candidates to anti-EGFR rechallenge.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Written informed consent to molecular analyses.
* Histologically proven diagnosis of CRC.
* At least one measurable lesion according to RECIST1.1
* ECOG PS ≤ 1.
* mCRC previously treated for metastatic disease with, or not considered candidates for, fluoropyrimidine, oxaliplatin, irinotecan and anti-angiogenic monoclonal antibody (bevacizumab or aflibercept).
* RAS (codons 12, 13, 59, 61, 117 and 146 of KRAS and NRAS genes) and BRAF (V600E mutation) wt status of primary CRC or related metastasis (local laboratory assessment).
* Previous first-line anti-EGFR-containing therapy producing at least a partial response or a stable disease ≥ 6 months.
* At least 4 months elapsed between the end of first-line anti-EGFR administration and screening.
* At least one line of therapy between the end of first-line anti-EGFR administration and screening.
* Availability of plasma sample for liquid biopsy within 28 days prior enrolment.
* RAS (codons 12, 13, 59, 61, 117 and 146 of KRAS and NRAS genes) and BRAF (V600E mutation) wt status of ct-DNA at screening (central laboratory assessment by means of IdyllaTM ctKRAS-NRAS-BRAF Mutation Test).
* Written informed consent to study treatment and procedures.
* Life expectancy of at least 12 weeks.
* Availability of archival tumour tissue (primary tumour and metastases or at least one of the two) for biomarker analysis.
* Availability of biological samples for translational molecular analyses.
* Neutrophils ≥1.5 x 109/L, Platelets ≥100 x 109/L, Hgb ≥ 9 g/dl.
* Total bilirubin ≤ 1.5 fold the upper-normal limits (UNL), ASAT (SGOT) and/or ALAT (SGPT) ≤ 2.5 x UNL (or <5 x UNL in the case of liver metastases), alkaline phosphatase ≤ 2.5 x UNL (or <5 x UNL in case of liver metastases).
* Creatinine clearance ≥ 50 mL/min or serum creatinine ≤1.5 x UNL.
* Women of childbearing potential must have a negative blood pregnancy test at the baseline visit. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 months, are surgically sterile, or are sexually inactive A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
* Subjects and their partners must be willing to avoid pregnancy during the trial and until 8 weeks after the last trial treatment. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception as approved by the investigator (barrier contraceptive measure or oral contraception).
* Will and ability to comply with the protocol.

Exclusion Criteria:

* Previous treatment with regorafenib.
* Radiotherapy to any site within 4 weeks before the study.
* Untreated brain metastases or spinal cord compression or primary brain tumours.
* Evidence of bleeding diathesis or coagulopathy.
* Uncontrolled hypertension and prior history of hypertensive crisis or hypertensive encephalopathy.
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication.
* Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of study enrolment.
* Any previous venous thromboembolism ≥ NCI CTCAE Grade 4.
* History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to the first study treatment.
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ.
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication.
* Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs.
* Any concomitant drugs contraindicated for use with the trial drugs according to the product information of the pharmaceutical companies.
* Diagnosis of interstitial pneumonitis or pulmonary fibrosis.
* Active uncontrolled infections or other clinically relevant concomitant illness contraindicating administration of panitumumab and regorafenib.
* Treatment with any investigational drug within 30 days prior to enrolment or 2 investigational agent half-lives (whichever is longer).
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Sexually active males and females (of childbearing potential) unwilling to practice contraception (barrier contraceptive measure or oral contraception) during the study and until 8 weeks after the last trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 30 months
  time from randomization to the date of death due to any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.

SECONDARY OUTCOMES:
Overall Toxicity Rate | 24 months
  percentage of patients, relative to the total of enrolled subjects, experiencing any adverse event, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during panitumumab and regorafenib
G3/4 Toxicity Rate | 24 months
  the percentage of patients, relative to the total of enrolled subjects, experiencing a specific adverse event of grade 3/4, according to National Cancer Institute Common Toxicity Criteria (version 5.0), during panitumumab and regorafenib.
1st-Progression free survival | 21 months
  time from randomization to the first documentation of objective disease progression or death due to any cause, whichever occurs first.
2nd-Progression free survival | 24 months
  the time from the beginning of the second-line study treatment to the documentation of objective disease progression according to RECIST 1.1 criteria or death due to any cause, whichever occurs first
Time to Failure of strategy | 24 months
  the time from randomization till the first of any of the following events: a) death; b) disease progression according to RECIST 1.1 criteria on any treatment given after 1st progression
Objective Response Rate | 24 months
  the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria, during panitumumab and regorafenib.

CONTACTS AND LOCATIONS:
Locations (1):
- U.O. Oncologia 2 Universitaria, Pisa, PI, Italy

IPD SHARING:
Plan to Share IPD: No